CLINICAL TRIAL: NCT00597467
Title: An Open-Labeled, Multi-Center, Randomized Investigation of the VISA (Comfilcon A) Silicone Hydrogel Soft (Hydrophilic) Contact Lens for Use in a 7 Day Extended Wear Regimen
Brief Title: Study of Soft Contact Lens Use With 7 Day Extended Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVI060105
Record Dates: First submitted 2007-12-27; First posted 2008-01-18 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Ametropia
Keywords: myopia; hyperopia; extended wear; ametropia
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test Contact Lenses (Experimental): VISA (comfilcon A) Silicone Hydrogel Soft contact lens
  Interventions: Device: VISA (comfilcon A) Silicone Hydrogel Soft contact lens
- Control Contact Lenses (Active Comparator): Acuvue 2 Soft Contact Lens
  Interventions: Device: Acuvue 2 Soft Contact Lens

INTERVENTIONS:
Device: VISA (comfilcon A) Silicone Hydrogel Soft contact lens — Test device
  Other Names: Biofinity (comfilcon A)
  Arms: Test Contact Lenses
Device: Acuvue 2 Soft Contact Lens — Control device
  Arms: Control Contact Lenses

SUMMARY:
To compare the safety and efficacy of the CVI silicone-hydrogel lens worn on an extended wear basis for a period of up to 7 days and 6 nights with the Acuvue 2 soft contact lenses.

DETAILED DESCRIPTION:
To compare the safety and efficacy of the CVI silicone-hydrogel lens worn on an extended wear basis for a period of up to 7 days and 6 nights with the Acuvue 2 soft contact lenses in this open-labeled randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age as of the date of evaluation.
2. Require lens powers between -0.50 and -6.00 diopters sphere with no more than 1.00 diopter of refractive astigmatism and be willing to wear lenses in both eyes.
3. Be correctable to visual acuities of at least 20/25 in each eye with spectacles.
4. Be in good general health, based on his/her knowledge.
5. Be able and willing to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
6. Possess wearable and visually functional eyeglasses.

Exclusion Criteria:

1. Previously unsuccessful with contact lens wear.
2. Rigid gas permeable contact lens wear within the past 12 months.
3. Previous refractive surgery; current or previous orthokeratology treatment.
4. Subject is wearing lenses in a modified monovision modality (multifocal lens in one eye). NOTE: subjects may not wear monovision lenses at any time during the study unless they are wearing spherical monovision lenses prior to enrollment.
5. Aphakia, keratoconus or an irregular cornea.
6. A known history of corneal hypoesthesia
7. Clinically significant (grade 3 or 4) anterior segment abnormalities or any infection of the eye, lids, or associated structures.
8. Ocular or systemic disease or need for medication which might interfere with contact lens wear. i.e., Sjögren's syndrome, type II diabetes, etc.
9. Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

   * History of corneal ulcer, corneal infiltrates or fungal infections.
   * Pterygium, pinguecula or corneal scars within the visual axis
   * Pathological dry eye or associated findings (examples: Sjögren's syndrome, lupus erythematosus, sclerodermia)
   * Neovascularization or ghost vessels > 1mm in from the limbus
   * Seborrheic eczema, seborrheic conjunctivitis
   * History of papillary conjunctivitis greater than Grade 2 (Mild)
   * Anterior uveitis or iritis (past or present)
10. Known sensitivity to the care systems used in this study.
11. Poor personal hygiene
12. Current pregnancy or is lactating (to the best of the subject's knowledge) or subject is planning pregnancy within the next 13 months.
13. Any active participation in another clinical study within 30 days prior to this study.
14. Subject is a member, relative or household member of the office staff, including the investigator(s).

Subjects must read, indicate understanding of, and sign the Informed Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Frequency of serious and significant AEs | 1 Year
  Frequency of serious and significant AEs defined as a composite of infiltrates of higher than grade 2 and/or infiltrates with any overlying staining, peripheral ulcer, and loss of two or more lines of visual acuity at any time during the trial

SECONDARY OUTCOMES:
Contact Lens Visual Acuity | 1 Year
  Contact lens visual acuity was assessed using LogMAR

CONTACTS AND LOCATIONS:
Overall Officials: William Gleason, OD, Study Director — FRS
Locations (23):
- United States (23):
  - La Mesa Vision Care Center, La Mesa, California
  - (Private Practice), San Diego, California
  - Drs. Cook, Reeder and Associates, San Diego, California
  - (Private Practice), Santa Monica, California
  - Eye Care Associates, P.C., Fort Collins, Colorado
  - Eola Eyes, Orlando, Florida
  - (Private Practice), Honolulu, Hawaii
  - Kato & Shoji Optometrists, Honolulu, Hawaii
  - Eye Care Associates of Hawaii, Waipahu, Hawaii
  - Davis Eyecare Associates, Oak Lawn, Illinois
  - (Private Practice), Andover, Massachusetts
  - Vision Care Associates, East Lansing, Michigan
  - The Koetting Associates Inc., St Louis, Missouri
  - Concord Ophthalmological Associates, Concord, New Hampshire
  - Place Optical Company Inc, Le Roy, New York
  - Quinn Quinn & Associates, Athens, Ohio
  - Western Reserve Vision Care, Beachwood, Ohio
  - Ohio State University, Columbus, Ohio
  - Professional Eye Care Associates, Columbus, Ohio
  - Primary Eyecare Group, P.C., Brentwood, Tennessee
  - (Private Practice), Salt Lake City, Utah
  - Twin Lakes Vision, Federal Way, Washington
  - Snowy Range Vision Center, Laramie, Wyoming